CLINICAL TRIAL: NCT05729035
Title: Predictive Value of Point of Care Ultrasound (POCUS) Versus Computerized Tomography (CT) in Diagnosis of Acute Dyspnea in Chronic Hemodialysis Patients.
Brief Title: POCUS VS CT in Diagnosis of Acute Dyspnea in Chronic Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Randa Ahmed Sarhan (Other)
Responsible Party: Sponsor-Investigator, Randa Ahmed Sarhan, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: POCUS VS CT chest
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Dyspnea; Chronic Renal Failure
MeSH Terms: conditions — Dyspnea; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: POCUS — Point of Care Ultrasound is complementary to a medical examination performed by primary care physicians
  Other Names: CT chest

SUMMARY:
Estimate the predictive value of POCUS in diagnosis of different causes of acute dyspnea in hemodialysis patients and compare between POCUS and CT in differentiation the causes of acute dyspnea in those population.

DETAILED DESCRIPTION:
Dyspnea is "a subjective experience of breathing discomfort that consists of qualitatively dis-tinct sensations that vary in intensity.Dyspnea is a common symptom both in general practice and in hospital emergency rooms. It has been reported that 7.4% of patients presenting to emergency rooms complain of dyspnea;among patients in general practice, 10% complain of dyspnea when walking on flat ground and 25% complain of dyspnea on more intense exertion, e.g., climbing stairs.Dyspnea is considered acute when it develops over hours to days.Acute breathlessness in haemodialysis patients can be caused by various conditions such as acute coronary syndrome, catheter-related infection, pneumonia and pericardial effusion, as well as a reaction to the dialyser or medication given during dialysis Hence, clinical acumen remains integral in evaluation of acute breathlessness in this group of patients. Point of Care Ultrasound is complementary to a medical examination performed by primary care physicians in conjunction to physical examination to investigate unclear findings. As such it is used to find and identify either the presence or absence of specific pathological results seen in your patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients maintained on regular hemodialysis equal to / more than 6 months admitted to emergency department and ICU of Internal Medicine Department from September 2021 to August 2022 presented by acute dyspnea.

Exclusion Criteria:

* • Age less than 18

  * Diagnosed chronic pulmonary disease.
  * Severe heart failure (NYHA class IV).
  * Active malignancy.
  * Pregnancy.
  * Hepatic Failure (Child B,C).
  * Comatosed Patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - All patients maintained on regular hemodialysis equal to / more than 6 months admitted to emergency department and ICU of Internal Medicine Department from September 2021 to August 2022 presented by acute dyspnea.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Compare between POCUS and CT in differentiation the causes of acute dyspnea in hemodialysis patients. | All patients maintained on regular hemodialysis equal to / more than 6 months admitted to emergency department and ICU of Internal Medicine Department from September 2021 to August 2022 presented by acute dyspnea
  Predictive value of Point of Care Ultrasound (POCUS) versus computerized tomography (CT) in Diagnosis of Acute Dyspnea in Chronic Hemodialysis Patients.

REFERENCES:
- [Background] Smallwood N, Dachsel M. Point-of-care ultrasound (POCUS): unnecessary gadgetry or evidence-based medicine? Clin Med (Lond). 2018 Jun;18(3):219-224. doi: 10.7861/clinmedicine.18-3-219. PMID 29858431
- [Background] Li L, Yong RJ, Kaye AD, Urman RD. Perioperative Point of Care Ultrasound (POCUS) for Anesthesiologists: an Overview. Curr Pain Headache Rep. 2020 Mar 21;24(5):20. doi: 10.1007/s11916-020-0847-0. PMID 32200432
- [Background] Rice JA, Brewer J, Speaks T, Choi C, Lahsaei P, Romito BT. The POCUS Consult: How Point of Care Ultrasound Helps Guide Medical Decision Making. Int J Gen Med. 2021 Dec 15;14:9789-9806. doi: 10.2147/IJGM.S339476. eCollection 2021. PMID 34938102